CLINICAL TRIAL: NCT05020626
Title: Modelling Tau Deposition and Distribution From Diffusion Tensor Imaging With Generative Adversarial Network for Alzheimer's Disease Diagnosis
Brief Title: Modelling Tau Distribution From DTI With Generative Adversarial Network for Alzheimer's Disease Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Other Study IDs: 2021.243
Record Dates: First submitted 2021-08-04; First posted 2021-08-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease Diagnosis
Keywords: Generative Adversarial Network; Tau; Diffusion Tensor Imaging
MeSH Terms: conditions — Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls
- Mild cognitive impairment
- AD dementia

SUMMARY:
The most significant impact of this project is to propose for the first time a novel generative adversarial network (GAN), as one kind of deep learning architecture, to automatically generate synthetic PET images reflecting tau deposition, from brain DTI images. If successful, this framework will become the most state-of-the-art approach to simulate the stereotypical pattern of intracerebral tau accumulation and distribution in vivo.

Synthetic tau-PET images via DTI, possessing overwhelming superiority in radiation-free, non-invasiveness and cost-effectiveness, will potentially serve as one of alternative modalities of PET in detecting tau-load and probably outperform PET on accessibility, generalizability, and availability in future, making it much more attractive in clinical application. A big conceptual shift may occur preferring a fire-new tau-PET simulated via DTI.

The DTI data-driven deep learning framework to be created in this project will constitute an accurate, robust, clinically applicable and explainable tool to efficiently categorize the subjects into tau-burden positive and tau-burden negative cases, which will undoubtedly contribute to both clinical and research activities.

ELIGIBILITY:
Inclusion Criteria:

* With the age of 55 years and above
* With brain MRI taken within ±6 months from the date of clinically confirmed diagnosis of AD, MCI or normal cognition.

Exclusion Criteria:

* AD with mixed dementia
* Non-AD dementia
* History of severe traumatic brain injury, severe depression, stroke, brain tumors, and incident major systemic illness

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The data will be collected from a public database, i.e, Alzheimer's Disease Nueroimaging Initiative (ADNI). According to their recruitment protocol at http://adni.loni.usc.edu/methods/documents/, the study enrolls men and women aged 55-90 years across MCI and mild AD dementia participant groups, and control normal aged 65 years with exceptions granted for minority participants.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural similarity index to measure the similarity between synthetic image and ground truth for 20% of data in testing set | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Background] Lane CA, Hardy J, Schott JM. Alzheimer's disease. Eur J Neurol. 2018 Jan;25(1):59-70. doi: 10.1111/ene.13439. Epub 2017 Oct 19. PMID 28872215
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Scheltens P, Blennow K, Breteler MM, de Strooper B, Frisoni GB, Salloway S, Van der Flier WM. Alzheimer's disease. Lancet. 2016 Jul 30;388(10043):505-17. doi: 10.1016/S0140-6736(15)01124-1. Epub 2016 Feb 24. PMID 26921134
- [Background] Hyman BT, Phelps CH, Beach TG, Bigio EH, Cairns NJ, Carrillo MC, Dickson DW, Duyckaerts C, Frosch MP, Masliah E, Mirra SS, Nelson PT, Schneider JA, Thal DR, Thies B, Trojanowski JQ, Vinters HV, Montine TJ. National Institute on Aging-Alzheimer's Association guidelines for the neuropathologic assessment of Alzheimer's disease. Alzheimers Dement. 2012 Jan;8(1):1-13. doi: 10.1016/j.jalz.2011.10.007. PMID 22265587
- [Background] Khan TK. An Algorithm for Preclinical Diagnosis of Alzheimer's Disease. Front Neurosci. 2018 Apr 30;12:275. doi: 10.3389/fnins.2018.00275. eCollection 2018. PMID 29760644
- [Background] Mito R, Raffelt D, Dhollander T, Vaughan DN, Tournier JD, Salvado O, Brodtmann A, Rowe CC, Villemagne VL, Connelly A. Fibre-specific white matter reductions in Alzheimer's disease and mild cognitive impairment. Brain. 2018 Mar 1;141(3):888-902. doi: 10.1093/brain/awx355. PMID 29309541
- [Background] Espay AJ, Vizcarra JA, Marsili L, Lang AE, Simon DK, Merola A, Josephs KA, Fasano A, Morgante F, Savica R, Greenamyre JT, Cambi F, Yamasaki TR, Tanner CM, Gan-Or Z, Litvan I, Mata IF, Zabetian CP, Brundin P, Fernandez HH, Standaert DG, Kauffman MA, Schwarzschild MA, Sardi SP, Sherer T, Perry G, Leverenz JB. Revisiting protein aggregation as pathogenic in sporadic Parkinson and Alzheimer diseases. Neurology. 2019 Feb 12;92(7):329-337. doi: 10.1212/WNL.0000000000006926. PMID 30745444
- [Background] Baker JE, Lim YY, Pietrzak RH, Hassenstab J, Snyder PJ, Masters CL, Maruff P. Cognitive impairment and decline in cognitively normal older adults with high amyloid-beta: A meta-analysis. Alzheimers Dement (Amst). 2016 Oct 18;6:108-121. doi: 10.1016/j.dadm.2016.09.002. eCollection 2017. PMID 28239636
- [Background] Hedden T, Oh H, Younger AP, Patel TA. Meta-analysis of amyloid-cognition relations in cognitively normal older adults. Neurology. 2013 Apr 2;80(14):1341-8. doi: 10.1212/WNL.0b013e31828ab35d. PMID 23547267
- [Background] Gordon BA, McCullough A, Mishra S, Blazey TM, Su Y, Christensen J, Dincer A, Jackson K, Hornbeck RC, Morris JC, Ances BM, Benzinger TLS. Cross-sectional and longitudinal atrophy is preferentially associated with tau rather than amyloid beta positron emission tomography pathology. Alzheimers Dement (Amst). 2018 Mar 6;10:245-252. doi: 10.1016/j.dadm.2018.02.003. eCollection 2018. PMID 29780869
- [Background] Xia C, Makaretz SJ, Caso C, McGinnis S, Gomperts SN, Sepulcre J, Gomez-Isla T, Hyman BT, Schultz A, Vasdev N, Johnson KA, Dickerson BC. Association of In Vivo [18F]AV-1451 Tau PET Imaging Results With Cortical Atrophy and Symptoms in Typical and Atypical Alzheimer Disease. JAMA Neurol. 2017 Apr 1;74(4):427-436. doi: 10.1001/jamaneurol.2016.5755. PMID 28241163
- [Background] Bejanin A, Schonhaut DR, La Joie R, Kramer JH, Baker SL, Sosa N, Ayakta N, Cantwell A, Janabi M, Lauriola M, O'Neil JP, Gorno-Tempini ML, Miller ZA, Rosen HJ, Miller BL, Jagust WJ, Rabinovici GD. Tau pathology and neurodegeneration contribute to cognitive impairment in Alzheimer's disease. Brain. 2017 Dec 1;140(12):3286-3300. doi: 10.1093/brain/awx243. PMID 29053874
- [Background] Sepulcre J, Grothe MJ, d'Oleire Uquillas F, Ortiz-Teran L, Diez I, Yang HS, Jacobs HIL, Hanseeuw BJ, Li Q, El-Fakhri G, Sperling RA, Johnson KA. Neurogenetic contributions to amyloid beta and tau spreading in the human cortex. Nat Med. 2018 Dec;24(12):1910-1918. doi: 10.1038/s41591-018-0206-4. Epub 2018 Oct 29. PMID 30374196
- [Background] Ossenkoppele R, Schonhaut DR, Scholl M, Lockhart SN, Ayakta N, Baker SL, O'Neil JP, Janabi M, Lazaris A, Cantwell A, Vogel J, Santos M, Miller ZA, Bettcher BM, Vossel KA, Kramer JH, Gorno-Tempini ML, Miller BL, Jagust WJ, Rabinovici GD. Tau PET patterns mirror clinical and neuroanatomical variability in Alzheimer's disease. Brain. 2016 May;139(Pt 5):1551-67. doi: 10.1093/brain/aww027. Epub 2016 Mar 8. PMID 26962052
- [Background] VandeVrede L, Boxer AL, Polydoro M. Targeting tau: Clinical trials and novel therapeutic approaches. Neurosci Lett. 2020 Jul 13;731:134919. doi: 10.1016/j.neulet.2020.134919. Epub 2020 May 4. PMID 32380145
- [Background] Lashley T, Schott JM, Weston P, Murray CE, Wellington H, Keshavan A, Foti SC, Foiani M, Toombs J, Rohrer JD, Heslegrave A, Zetterberg H. Molecular biomarkers of Alzheimer's disease: progress and prospects. Dis Model Mech. 2018 May 8;11(5):dmm031781. doi: 10.1242/dmm.031781. PMID 29739861
- [Background] Jacobs HIL, Hedden T, Schultz AP, Sepulcre J, Perea RD, Amariglio RE, Papp KV, Rentz DM, Sperling RA, Johnson KA. Structural tract alterations predict downstream tau accumulation in amyloid-positive older individuals. Nat Neurosci. 2018 Mar;21(3):424-431. doi: 10.1038/s41593-018-0070-z. Epub 2018 Feb 5. PMID 29403032
- [Background] Wen Q, Risacher SL, Xie L, Li J, Harezlak J, Farlow MR, Unverzagt FW, Gao S, Apostolova LG, Saykin AJ, Wu YC. Tau-related white-matter alterations along spatially selective pathways. Neuroimage. 2021 Feb 1;226:117560. doi: 10.1016/j.neuroimage.2020.117560. Epub 2020 Nov 12. PMID 33189932
- [Background] Braak H, Braak E. Frequency of stages of Alzheimer-related lesions in different age categories. Neurobiol Aging. 1997 Jul-Aug;18(4):351-7. doi: 10.1016/s0197-4580(97)00056-0. PMID 9330961
- [Background] Braak H, Thal DR, Ghebremedhin E, Del Tredici K. Stages of the pathologic process in Alzheimer disease: age categories from 1 to 100 years. J Neuropathol Exp Neurol. 2011 Nov;70(11):960-9. doi: 10.1097/NEN.0b013e318232a379. PMID 22002422
- [Background] Grinberg LT, Rub U, Ferretti RE, Nitrini R, Farfel JM, Polichiso L, Gierga K, Jacob-Filho W, Heinsen H; Brazilian Brain Bank Study Group. The dorsal raphe nucleus shows phospho-tau neurofibrillary changes before the transentorhinal region in Alzheimer's disease. A precocious onset? Neuropathol Appl Neurobiol. 2009 Aug;35(4):406-16. doi: 10.1111/j.1365-2990.2009.00997.x. PMID 19508444
- [Background] Olsson B, Lautner R, Andreasson U, Ohrfelt A, Portelius E, Bjerke M, Holtta M, Rosen C, Olsson C, Strobel G, Wu E, Dakin K, Petzold M, Blennow K, Zetterberg H. CSF and blood biomarkers for the diagnosis of Alzheimer's disease: a systematic review and meta-analysis. Lancet Neurol. 2016 Jun;15(7):673-684. doi: 10.1016/S1474-4422(16)00070-3. Epub 2016 Apr 8. PMID 27068280
- [Background] Hameed S, Fuh JL, Senanarong V, Ebenezer EGM, Looi I, Dominguez JC, Park KW, Karanam AK, Simon O. Role of Fluid Biomarkers and PET Imaging in Early Diagnosis and its Clinical Implication in the Management of Alzheimer's Disease. J Alzheimers Dis Rep. 2020 Feb 12;4(1):21-37. doi: 10.3233/ADR-190143. PMID 32206755
- [Background] Hampel H, O'Bryant SE, Molinuevo JL, Zetterberg H, Masters CL, Lista S, Kiddle SJ, Batrla R, Blennow K. Blood-based biomarkers for Alzheimer disease: mapping the road to the clinic. Nat Rev Neurol. 2018 Nov;14(11):639-652. doi: 10.1038/s41582-018-0079-7. PMID 30297701
- [Background] de Almeida SM, Shumaker SD, LeBlanc SK, Delaney P, Marquie-Beck J, Ueland S, Alexander T, Ellis RJ. Incidence of post-dural puncture headache in research volunteers. Headache. 2011 Nov-Dec;51(10):1503-10. doi: 10.1111/j.1526-4610.2011.01959.x. Epub 2011 Jul 28. PMID 21797856
- [Background] Caso F, Agosta F, Filippi M. Insights into White Matter Damage in Alzheimer's Disease: From Postmortem to in vivo Diffusion Tensor MRI Studies. Neurodegener Dis. 2016;16(1-2):26-33. doi: 10.1159/000441422. Epub 2015 Dec 1. PMID 26618812
- [Background] Kantarci K, Murray ME, Schwarz CG, Reid RI, Przybelski SA, Lesnick T, Zuk SM, Raman MR, Senjem ML, Gunter JL, Boeve BF, Knopman DS, Parisi JE, Petersen RC, Jack CR Jr, Dickson DW. White-matter integrity on DTI and the pathologic staging of Alzheimer's disease. Neurobiol Aging. 2017 Aug;56:172-179. doi: 10.1016/j.neurobiolaging.2017.04.024. Epub 2017 May 4. PMID 28552181
- [Background] Oishi K, Mielke MM, Albert M, Lyketsos CG, Mori S. DTI analyses and clinical applications in Alzheimer's disease. J Alzheimers Dis. 2011;26 Suppl 3(Suppl 3):287-96. doi: 10.3233/JAD-2011-0007. PMID 21971468
- [Background] Tang X, Qin Y, Wu J, Zhang M, Zhu W, Miller MI. Shape and diffusion tensor imaging based integrative analysis of the hippocampus and the amygdala in Alzheimer's disease. Magn Reson Imaging. 2016 Oct;34(8):1087-99. doi: 10.1016/j.mri.2016.05.001. Epub 2016 May 20. PMID 27211255
- [Background] Mayo CD, Mazerolle EL, Ritchie L, Fisk JD, Gawryluk JR; Alzheimer's Disease Neuroimaging Initiative. Longitudinal changes in microstructural white matter metrics in Alzheimer's disease. Neuroimage Clin. 2016 Dec 16;13:330-338. doi: 10.1016/j.nicl.2016.12.012. eCollection 2017. PMID 28066707
- [Background] de la Monte SM. Quantitation of cerebral atrophy in preclinical and end-stage Alzheimer's disease. Ann Neurol. 1989 May;25(5):450-9. doi: 10.1002/ana.410250506. PMID 2774485